CLINICAL TRIAL: NCT02309320
Title: A Phase I/IIa Multicentre Study in Otherwise Healthy Infants and Toddlers Hospitalised For and Diagnosed With Respiratory Syncytial Virus Lower Respiratory Tract Infection, Consisting of an Open-label Lead-in Part Followed by a Double-blind, Placebo-controlled Part, to Evaluate the Safety, Tolerability and Clinical Activity of ALX-0171, Administered Via Inhalation, in Addition to Standard of Care.
Brief Title: A Multicentre Study in Otherwise Healthy Infants and Toddlers Hospitalised For and Diagnosed With RSV Lower Respiratory Tract Infection to Evaluate the Safety, Tolerability, and Clinical Activity of ALX-0171
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ablynx, a Sanofi company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALX0171-C104; 2014-002841-23 (EudraCT Number)
Record Dates: First submitted 2014-11-27; First posted 2014-12-05 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Respiratory Syncytial Virus Infection
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — gontivimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ALX-0171 (Experimental): Inhalation of ALX-0171 during 3 consecutive days
  Interventions: Biological: ALX-0171
- Placebo (Placebo Comparator): Inhalation of Placebo during 3 consecutive days
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: ALX-0171
  Arms: ALX-0171
Other: Placebo
  Arms: Placebo

SUMMARY:
The primary objective of the study is to investigate the safety and tolerability of ALX-0171.

The secondary objectives are to evaluate the clinical effect of ALX-0171 and to explore the pharmacodynamics (PD) and the systemic pharmacokinetics (PK) of ALX-0171.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is otherwise healthy, but hospitalised for and clinically diagnosed with RSV LRTI (Lower Respiratory Tract Infection)
2. Subject has appearance of upper or lower respiratory tract infection symptoms that are likely related to RSV
3. Subject has a positive RSV diagnostic test
4. Others as defined in the protocol

Exclusion Criteria:

1. Subject has history of wheezing
2. Subject is known to have significant comorbidities
3. Subject is known to be immunocompromised
4. Subject is suspected of having a clinically relevant infection other than RSV
5. Others as defined in the protocol

Ages: 28 Days to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability as measured by the incidence of treatment emergent adverse events, clinical laboratory parameters and physical examination | 1 day before first dose to 14 days after first dose

SECONDARY OUTCOMES:
Clinical activity as measured by the evaluation of the clinical response of the subjects | 1 day before first dose to 14 days after first dose
Exploratory Pharmacokinetics as measured by the concentration of ALX-0171 in serum | Day 3
Exploratory Pharmacodynamics as measured by the concentration of viral load in respiratory secretions and exploratory biomarkers in serum | 1 day before first dose to 14 days after first dose
Immunogenicity as measured by the concentration of anti-drug antibodies in serum | 1 day before first dose to 14 days after first dose

CONTACTS AND LOCATIONS:
Overall Officials: Ablynx Clinical Department, Study Director — Ablynx, a Sanofi company
Locations (59):
- Australia (4):
  - Investigator Site 4, Brisbane
  - Investigator Site 2, Randwick
  - Investigator Site 3, Tasmania
  - Investigator Site 1, Westmead
- Belgium (6):
  - Investigator Site 1, Antwerp
  - Investigator Site 6, Antwerp
  - Investigator Site 4, Brussels
  - Investigator Site 5, Brussels
  - Investigator Site 2, Ghent
  - Investigator Site 3, Leuven
- Bulgaria (4):
  - Investigator Site 4, Kozloduy
  - Investigator Site 1, Pleven
  - Investigator Site 2, Rousse
  - Investigator Site 3, Sevlievo
- Investigator Site, Tartu, Estonia
- Hungary (5):
  - Investigator Site 1, Budapest
  - Investigators Site 3, Budapest
  - Investigator Site 4, Budapest
  - Investigator Site 5, Budapest
  - Investigator Site 2, Szeged
- Israel (3):
  - Investigator Site 3, Beersheba
  - Investigator Site 2, Haifa
  - Investigator Site 1, Petah Tikva
- Latvia (3):
  - Investigator Site 3, Daugavpils
  - Investigator Site 2, Riga
  - Investigator Site 1, Valmiera
- Malaysia (4):
  - Investigator Site 2, Ipoh
  - Investigator Site 1, Kuala Lumpur
  - Investigator Site 3, Negeri Sembilan
  - Investigator Site 4, Pulau Pinang
- Philippines (3):
  - Investigator Site, City of Muntinlupa
  - Investigator Site, Manila
  - Investigator Site, Quezon City
- Poland (3):
  - Investigator Site 3, Bydgoszcz
  - Investigator Site 2, Lodz
  - Investigator Site 1, Trzebnica
- Slovakia (7):
  - Investigator Site 5, Banská Bystrica
  - Investigator Site 3, Bratislava
  - Investigator Site 2, Košice
  - Investigator Site 6, Levice
  - Investigator Site 7, Liptovský Mikuláš
  - Investigator Site 1, Martin
  - Investigator Site 4, Poprad
- Spain (8):
  - Investigator Site 5, Barcelona
  - Investigator Site 2, Barcelona
  - Investigator Site 4, Girona
  - Investigator Site 3, Madrid
  - Investigator Site 7, Málaga
  - Investigator Site 6, Murcia
  - Investigator Site 1, Santiago de Compostela
  - Investigator Site 8, Seville
- Thailand (2):
  - Investigator Site 2, Chiang Mai
  - Investigator Site, Khon Kaen
- United Kingdom (6):
  - Investigator Site 2, City of Edinburgh
  - Investigator Site 4, Kent
  - Investigator Site 5, Liverpool
  - Investigator Site 6, Nottingham
  - Investigator Site 1, Oxford
  - Investigator Site 3, Tooting